CLINICAL TRIAL: NCT05927285
Title: Effect on Kidney Function Recovery Guiding Decongestion With VExUS in Patients With Cardiorenal Syndrome 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, Jonathan Samuel Chavez Iñiguez, Dr., Hospital Civil de Guadalajara
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HCG/CEI-0836/22
Record Dates: First submitted 2023-06-12; First posted 2023-07-03 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Cardiorenal Syndrome; Acute Kidney Injury; Decompensated Heart Failure; Fluid Overload; Ultrasound Therapy; Complications
MeSH Terms: conditions — Cardio-Renal Syndrome; Acute Kidney Injury; Edema | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The control group is considered the conventional approach, where the treatment was guided by improvement in clinical data, imaging, or laboratory studies during the daily evaluation until categorized as decongested.
  The VExUS group was considered the intervention group, where in addition to all the above, the decision for decongestant treatment was guided by the VExUS score until reaching a score that VExUS considered noncongestive, which was grade 0.
Who Masked: Participant
Masking Description: Allocation was performed by the cardiology staff on a concealed opaque envelope until the beginning of the study. A double-blind, double dummy design was used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VeXUS group (Experimental): The VExUS group was considered the intervention group, where in addition to all the above, the decision for decongestant treatment was guided by the VExUS score until reaching a score that VExUS considered noncongestive, which was grade 0.
  Interventions: Diagnostic Test: Vexus
- Control group (Active Comparator): The control group is considered the conventional approach, where the treatment was guided by improvement in clinical data, imaging, or laboratory studies during the daily evaluation until categorized as decongested.
  Interventions: Other: Control group

INTERVENTIONS:
Diagnostic Test: Vexus — The VExUS group was considered the intervention group, where in addition to all the above, the decision for decongestant treatment was guided by the VExUS score until reaching a score that VExUS considered noncongestive, which was grade 0.
  Arms: VeXUS group
Other: Control group — The control group is considered the conventional approach, where the treatment was guided by improvement in clinical data, imaging, or laboratory studies during the daily evaluation until categorized as decongested
  Arms: Control group

SUMMARY:
During cardiorenal syndrome type 1 (CRS1) vascular congestion is the major contributor to worsening renal function, but promoting decongestion with routine clinical evaluation is ineffective in some patients. The venous evaluation by ultrasound (VExUS) may optimize its management when evaluating for improvement in kidney function and other metrics related to decongestion.

DETAILED DESCRIPTION:
Background: In cardiorenal syndrome type 1 (CRS1) vascular congestion is a common complication, the Venus Evaluation by Ultrasound System (VExUS) could guide decongestion effectively and thereby improve kidney function outcomes.

Methods: In this double-blind randomized clinical trial, patients with CRS1 were randomized to guide decongestion with VExUS compared to usual clinical evaluation. The primary and secondary endpoint was to assess kidney function recovery (KFR), days of hospitalization, mortality, changes in brain natriuretic peptide (BNP) and CA-125. Protocol register HCG/CEI-0836/22.

ELIGIBILITY:
Inclusion Criteria:

* Cardiorenal Syndrome type 1

Exclusion Criteria:

* kidney transplantation, chronic kidney disease (CKD) grade 4 or 5, dialysis and pregnancy. CKD was defined according to the KDIGO guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2022-03-20 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-02-26 (Actual)

PRIMARY OUTCOMES:
Kidney Function Recovery | from hospitalization to discharge, or date of death from any cause, whichever came first, assessed up to 90 days
  Assess Kidney Function Recovery evaluated as serum Creatinine return to baseline value

SECONDARY OUTCOMES:
vascular decongestion during hospitalization | from hospitalization to discharge, or date of death from any cause, whichever came first, assessed up to 90 days
  Decongestion was defined as the following criteria: absence of peripheral edema, absence of orthopnea, no jugular ingurgitation, decreased or absent dyspnea, >30% decrease in BNP, CA 125 <35 ug/dL, chest X-ray without evidence of congestion, and less than days of hospitalization, mortality, changes in brain natriuretic peptide (BNP) and CA-125

OTHER OUTCOMES:
Exploratory outcomes | 90 days
  days of hospitalization
survival | 90 days
  dead for any cause

CONTACTS AND LOCATIONS:
Locations (1):
- HCG, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: Yes
If researchers required we can share data
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 2 weeks

REFERENCES:
- [Result] Hatamizadeh P, Fonarow GC, Budoff MJ, Darabian S, Kovesdy CP, Kalantar-Zadeh K. Cardiorenal syndrome: pathophysiology and potential targets for clinical management. Nat Rev Nephrol. 2013 Feb;9(2):99-111. doi: 10.1038/nrneph.2012.279. Epub 2012 Dec 18. PMID 23247571
- [Result] Chavez-Iniguez JS, Sanchez-Villaseca SJ, Garcia-Macias LA. [Cardiorenal syndrome: classification, pathophysiology, diagnosis and management. Literature review]. Arch Cardiol Mex. 2022 Apr 4;92(2):253-263. doi: 10.24875/ACM.20000183. Spanish. PMID 34261129
- [Result] Vandenberghe W, Gevaert S, Kellum JA, Bagshaw SM, Peperstraete H, Herck I, Decruyenaere J, Hoste EA. Acute Kidney Injury in Cardiorenal Syndrome Type 1 Patients: A Systematic Review and Meta-Analysis. Cardiorenal Med. 2016 Feb;6(2):116-28. doi: 10.1159/000442300. Epub 2015 Dec 19. PMID 26989397
- [Result] Chavez-Iniguez JS, Ibarra-Estrada M, Sanchez-Villaseca S, Romero-Gonzalez G, Font-Yanez JJ, De la Torre-Quiroga A, de Quevedo AA, Romero-Munoz A, Maggiani-Aguilera P, Chavez-Alonso G, Gomez-Fregoso J, Garcia-Garcia G. The Effect in Renal Function and Vascular Decongestion in Type 1 Cardiorenal Syndrome Treated with Two Strategies of Diuretics, a Pilot Randomized Trial. BMC Nephrol. 2022 Jan 3;23(1):3. doi: 10.1186/s12882-021-02637-y. PMID 34979962
- [Result] Husain-Syed F, Grone HJ, Assmus B, Bauer P, Gall H, Seeger W, Ghofrani A, Ronco C, Birk HW. Congestive nephropathy: a neglected entity? Proposal for diagnostic criteria and future perspectives. ESC Heart Fail. 2021 Feb;8(1):183-203. doi: 10.1002/ehf2.13118. Epub 2020 Nov 30. PMID 33258308
- [Result] Rocha BML, Menezes Falcao L. Acute decompensated heart failure (ADHF): A comprehensive contemporary review on preventing early readmissions and postdischarge death. Int J Cardiol. 2016 Nov 15;223:1035-1044. doi: 10.1016/j.ijcard.2016.07.259. Epub 2016 Aug 3. PMID 27592046
- [Derived] Islas-Rodriguez JP, Miranda-Aquino T, Romero-Gonzalez G, Hernandez-Del Rio J, Camacho-Guerrero JR, Covarrubias-Villa S, Ivey-Miranda JB, Chavez-Iniguez JS. Effect on Kidney Function Recovery Guiding Decongestion with VExUS in Patients with Cardiorenal Syndrome 1: A Randomized Control Trial. Cardiorenal Med. 2024;14(1):1-11. doi: 10.1159/000535641. Epub 2023 Dec 7. PMID 38061346